CLINICAL TRIAL: NCT05578638
Title: A Randomized Prospective Clinical Study on the Effect of Aloe Vera Gel and Rosmery Oil for Skin Ulcer Protection in Orthopedic Wards
Brief Title: Comparing Aloe Vera Gel and Rosemary Oil in Pressure Injury Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, mohamed elsayed hamed elzeky, lecturer at medical surgical nursing, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mans u
Record Dates: First submitted 2022-10-03; First posted 2022-10-13 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- aloe Vera group (Experimental): 10 ml of the spray will be rubbed two times per day during the skin care on the areas at risk for PIs, including the patient's sacrum area, hip areas and heels area. This action will continue for 10 days
  Interventions: Combination Product: aloevera tropical application
- rosemary group (Experimental): 10 ml of the spray will be rubbed two times per day during the skin care on the areas at risk for PIs, including the patient's sacrum area, hip areas and heels area. This action will continue for 10 days
  Interventions: Combination Product: rosemary tropicalapplication
- aloe Vera rosemary compound (Experimental): 10 ml of the spray will be rubbed two times per day during the skin care on the areas at risk for PIs, including the patient's sacrum area, hip areas and heels area. This action will continue for 10 days
  Interventions: Combination Product: Aloe Vera rosemary tropical application
- control group (No Intervention)

INTERVENTIONS:
Combination Product: Aloe Vera rosemary tropical application — 10 ml of the Aloe Vera rosemary spray will be rubbed two times per day during the skin care on the areas at risk for PIs, including the patient's sacrum area, hip areas and heels area. This action will continue for 10 days
  Arms: aloe Vera rosemary compound
Combination Product: aloevera tropical application — 10 ml of the Aloe Vera spray will be rubbed two times per day during the skin care on the areas at risk for PIs, including the patient's sacrum area, hip areas and heels area. This action will continue for 10 days
  Arms: aloe Vera group
Combination Product: rosemary tropicalapplication — 10 ml of the rosemary spray will be rubbed two times per day during the skin care on the areas at risk for PIs, including the patient's sacrum area, hip areas and heels area. This action will continue for 10 days
  Arms: rosemary group

SUMMARY:
Most patients admitted to the orthopedic ward are at risk of developing pressure ulcers. Today, the tendency to use medicinal herbs in pressure ulcer treatment has increased due to the variety of effective compounds and their fewer side effects.

DETAILED DESCRIPTION:
Aloe Vera is medicinal plant that has been used to treat skin problems since 1500 BC Many studies have shown that using Aloe Vera to treat various wounds such as psoriasis, mouth ulcers, diabetic ulcers herpes and bed sores has had positive effects. in addition, Rosemary has therapeutic properties and has been used in the folk medicine, pharmaceutical, and cosmetics industries, mainly for its antioxidant, anti-inflammatory and vasodilatation properties, which are attributed to the presence of carnosol/carnosic and ursolic acids. Besides it therapeutic uses, rosemary has potential applications in cosmetic formulations and in the treatment of pathological and non-pathological conditions, such as cellulite, alopecia, ultraviolet damage, and aging.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in research, lack of skin diseases (such as psoriasis, fungal illness, freckles), patients that are at risk of moderate to severe bedsores according to nursing diagnosis and Braden scoring tool and scored less than 13-14; the absence of PI on admission; the probability of length of stay should be above 10 days

Exclusion Criteria:

* a decrease in hemoglobin levels during the study to lower than 12 in men and less than 10 mg/dl in women, anemia, hyperthermia during the study and sensitivity to Aloe Vera or Rosemary.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
incidence of stage 1 pressure ulcers | Before applying sprays, Patients will be evaluated by pairs of observers (trained nurse and specialist) at 9:00 am for the presence of PIs at third day, after intervention
  The NPUAP scale is staging system since 1989 as one of the most widely used classification systems for the PI that describes the depth of the wound caused by PIs. In accordance with the panel, the PIs are divided into the original 4 stages and adding 2 stages on deep tissue injury and unstageable PIs. In this work, skin redness without discoloration by finger pressure in area of interest was considered as PIs stage I
incidence of stage 1 pressure ulcers | Before applying sprays, Patients will be evaluated by pairs of observers (trained nurse and specialist) at 9:00 am for the presence of PIs at seventh day, after intervention
  The NPUAP scale is staging system since 1989 as one of the most widely used classification systems for the PI that describes the depth of the wound caused by PIs. In accordance with the panel, the PIs are divided into the original 4 stages and adding 2 stages on deep tissue injury and unstageable PIs. In this work, skin redness without discoloration by finger pressure in area of interest was considered as PIs stage I
incidence of stage 1 pressure ulcers | Before applying sprays, Patients will be evaluated by pairs of observers (trained nurse and specialist) at 9:00 am for the presence of PIs at the tenth day, after intervention
  The NPUAP scale is staging system since 1989 as one of the most widely used classification systems for the PI that describes the depth of the wound caused by PIs. In accordance with the panel, the PIs are divided into the original 4 stages and adding 2 stages on deep tissue injury and unstageable PIs. In this work, skin redness without discoloration by finger pressure in area of interest was considered as PIs stage I
change in skin temperature at pressure points | will be measured at baseline and at the end of the study (after 10 days)
  Skin temperature will be measured using infrared thermometer
change in pain level at pressure points | will be measured at baseline and at the end of the study (after 10 days)
  pain will be measured using 0-10 visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No